CLINICAL TRIAL: NCT05715216
Title: EON: A Single-arm Phase II Study of Etigilimab (OMP-313M32) in Combination With Checkpoint Inhibition (Nivolumab) in Patients With Platinum-resistant, Recurrent Epithelial Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0896; NCI-2023-00827 (Other: NCI-CTRP Clinical Trials Registry); 2021-0511 (Registry Identifier: Clinical Trials Gov); NCT05026606 (obsolete NCT alias)
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etigilimab plus Nivolumab (Experimental): Participants will receive the study drugs on Days 1 and 15 of each study cycle,Cycle 1, Participants will receive the drugs on separate days (etigilimab on Day 1 and nivolumab on Day 2). Starting with Cycle 2, you will receive both drugs on Day 1 (separated by 2 hours).
  Interventions: Drug: Nivolumab; Drug: Etigilimab

INTERVENTIONS:
Drug: Nivolumab — Given by IV (vein)
  Other Names: BMS-936558; Opdivo
Drug: Etigilimab — Given by IV (vein)

SUMMARY:
To learn if adding etigilimab to nivolumab therapy can help to control clear cell ovarian, fallopian tube, and primary peritoneal cancers that are resistant to platinum-based therapy

DETAILED DESCRIPTION:
Primary Objectives:

1. To estimate the objective response rate of the combination of etigilimab and nivolumab in patients with platinum resistant clear cell ovarian cancer.
2. To evaluate the toxicity of the combination of etigilimab and nivolumab in patients with platinum resistant clear cell ovarian cancer.

Secondary Objectives:

1. To determine PFS of the combination of etigilimab and nivolumab in patients with platinum resistant clear cell ovarian cancer.
2. To estimate the disease control rate of the combination of etigilimab and nivolumab in patients with platinum resistant clear cell ovarian cancer.
3. To investigate molecular and immunological changes associated with the combination of TIGIT and PD-1 inhibition; specifically to describe changes in T cell populations (including but not limited to CD3, CD8, CD4, FOXP3) and cell proliferation, as well as report changes in the proportion of macrophage phenotypes M1 and M2 (with phenotypic markers potentially including arginase1, CD11b, PDL-1, and CD206)
4. To determine feasibility of interrogating the gut microbial signatures and dietary patterns in an ovarian cancer cohort.
5. Identify components and determinants of the gut microbiome that could modulate toxicity or provide a signature of excellent or poor response to cancer immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be assessed within 28 days of starting study treatment:

1. Ability to provide signed informed consent.
2. Age ≥ 18 years at time of study entry.
3. Willingness and ability to comply with the protocol for the duration of the study including undergoing treatment, biopsy, and scheduled visits and examinations including follow up.
4. Histology showing recurrent clear cell ovarian, peritoneal, or fallopian tube cancer.
5. Platinum resistant or refractory disease as defined by progression of disease on a platinum- containing regimen or recurrence of disease within 180 days of previous platinum treatment.

Have measurable disease based on modified RECIST 1.1. For the purposes of this study measurable disease is defined at least one "target lesion" that can be accurately measured in at least one dimension (longest dimension to be recorded). Each target lesion must be >20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >10 mm when measured by spiral CT. The target lesion must be distinct from other tumor areas selected for pre-treatment biopsies. Pre- treatment imaging must be performed within 4 weeks of starting therapy. 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 8. Adequate normal organ and marrow function as defined below.

1. Hemoglobin ≥9.0 g/dL.
2. Absolute neutrophil count (ANC) > 1500/mm3.
3. Platelet count ≥100 x 109/L (>75,000/mm3).
4. Serum bilirubin ≤1.5 x ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
5. AST (SGOT)/ALT (SGPT) ≤2.5 x ULN unless liver metastases are present, in which case it must be

   * 5x ULN.
6. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: Creatinine CL (mL/min)

   * Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL) 9. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients.

Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

1. Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post- menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy). 10. Has primary central nervous system (CNS) malignancy or known unrelated/active CNS metastases and/or carcinomatous meningitis.

<!-- -->

1. Subjects with previously treated, asymptomatic brain metastases may participate provided they meet the following criteria: clinically stable for at least 4 weeks and have no evidence of new or enlarging brain metastases and are off steroids 14 days prior to dosing with study medication. Stable brain metastases by this definition should be established prior to the first dose of study drug.
2. Subjects with asymptomatic brain metastases (ie, no neurological symptoms, no requirements for corticosteroids, and no lesion >1.5 cm) may participate but will require regular imaging of the brain as a site of disease.
3. Subjects with CNS symptoms should undergo a computed tomography (CT) scan or magnetic resonance imaging (MRI) of the brain to exclude new or progressive brain metastases. Spinal cord metastasis is acceptable. However, subjects with spinal cord compression must be excluded.

Exclusion Criteria:

Exclusion criteria will be assessed within 28 days of starting study treatment and is listed below.

1. Participation in another clinical study with an investigational product during the last 28 days.
2. Prior treatment with CD137 agonists, anti-TIGIT antibody, anti-CTLA-4 or anti-PDL1/PD1 antibodies.
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
4. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤28 days or 5 half-lives, whichever is shorter, prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by study sponsors and the investigator.
5. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the primary investigator.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with investigational therapy may be included only after consultation with the primary investigator.
6. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.
7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note:

   Local surgery of isolated lesions for palliative intent is acceptable.
8. History of allogenic organ transplantation.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criteria.

   a. Patients with vitiligo or alopecia. b. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.

   c. Any chronic skin condition that does not require systemic therapy. d. Patients without active disease in the last 5 years may be included but only after consultation with the primary investigator. e. Patients with celiac disease controlled by diet alone.
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
11. Any medical, social, or psychological condition that would interfere with evaluation of study treatment or interpretation of patient safety or study results.
12. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. History of another primary malignancy except for the following histories.

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.
14. History of leptomeningeal carcinomatosis.
15. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have a MRI (preferred) or CT each preferably with intravenous (IV) contrast of the brain prior to study entry.
16. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of trial therapies. Listed below are the exceptions to this criterion.

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP.
19. Female patients who are pregnant or breastfeeding or of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of Nivolumab/Etigilimab combination therapy.
20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
21. Unresolved partial or complete small or large bowel obstruction.
22. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org